CLINICAL TRIAL: NCT00105092
Title: A Phase II Evaluation of Oral Enzastaurin HCl in Second-and Third- Line Treatment of Patients With Non-Small Cell Lung Cancer
Brief Title: Enzastaurin as Second and Third-Line Treatment for Non-Small Cell Lung Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8670; H6Q-MC-JCAQ
Record Dates: First submitted 2005-03-04; First posted 2005-03-07 (Estimated); Last update posted 2007-05-01 (Estimated); Status verified 2007-04

CONDITIONS: Non-Small-Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — enzastaurin

INTERVENTIONS:
Drug: Enzastaurin HCL

SUMMARY:
Enzastaurin given daily to patients with non-small cell lung cancer who have failed at least one prior therapy.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old
* Must have been diagnosed with advanced or metastatic non-small cell lung cancer
* Must be able to visit the doctor's office every 28 days for 6 months or longer.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Have other significant medical problems as determined by your physician
* Are unable to swallow tablets
* Have a history of significant heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-03; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To estimate the rate of progression-free survival at 6 months for patients receiving oral enzastaurin with NSCLC who are eligible for second-or third-line therapy

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of enzastaurin using sparse sampling methodology in this population
To assess the QTc interval at anticipated steady state levels of enzastaurin (centrally collected 12-lead ECG on Day 1 of Cycle 2)
To estimate the objective response rate (complete response [CR] and partial response [PR])
To estimate time-to-event variables, such as overall survival time, duration of overall response (up to 1 year), and duration of stable disease (up to 1 year)
To evaluate the safety of enzastaurin in this patient population
To assess PKCb expression by immunohistochemistry in readily available tumors from patients
To evaluate enzastaurin's effect on patients' symptoms, functioning, and health-related quality of life using validated patient questionnaires
To explore biomarkers relevant to tumor progression and PKCb signaling

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Houston, Texas

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com